CLINICAL TRIAL: NCT05030610
Title: Treating Depression in Autistic Adults: A Feasibility Trial of an Adapted Behavioral Activation Program
Brief Title: Adaptation of a Behavioral Activation Treatment to Treat Depression in Autistic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Governor's Council for Medical Research and Treatment of Autism (Unknown)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Associate Professor; Karmazin & Lillard Chair in Adult Autism, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001254
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder; Depression; Depressive Symptoms
Keywords: behavioral activation
MeSH Terms: conditions — Autism Spectrum Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants, along with a support person, will complete 12 weekly sessions of the BeatIt-ASD intervention. The support person will complete an initial session before commencement of the 12 weekly sessions.
  Interventions: Behavioral: BeatIt-ASD

INTERVENTIONS:
Behavioral: BeatIt-ASD — BeatIt-ASD, designed to be implemented with autistic individuals, is an adaptation of BeatIt. The intervention aims to improve mood and decrease depressive symptoms through an increase in meaningful engagement in recreational, domestic, and social/leisure activities.

SUMMARY:
The present study aims to adapt and evaluate the feasibility of the BeatIt behavioral activation intervention for people with intellectual disabilities and low mood to be implemented with autistic individuals, with and without intellectual disabilities.

DETAILED DESCRIPTION:
The study has two specific aims:

1. Adapt BeatIt materials for use with autistic adults with and without Intellectual Disability (ID). Focus groups engaging key stakeholders will inform the adaptation of BeatIt for autistic adults (i.e., BeatIt-ASD). A stakeholder advisory team will provide input through the duration of the study.
2. Evaluate the feasibility, acceptability, and preliminary efficacy of BeatIt-ASD for autistic adults. This includes examining if the data demonstrate the feasibility and acceptability of the BeatIt-ASD program for autistic adults and provide preliminary evidence for behavioral change (i.e., increased engagement in meaningful activities and reduced depressive symptoms).

Data will demonstrate the feasibility and acceptability of the adapted BeatIt intervention for autistic adults and provide preliminary evidence for reduction of depression symptoms via regulation of routines and achievement of meaningful goals.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of Autism Spectrum Disorders (ASD)
2. Have a best estimate diagnosis of clinically significant depressive symptoms by the study team. This will be based on DSM-5 criteria or DM-ID (Diagnostic Manual - Intellectual Disability).
3. Have a support person willing to participate
4. Live in New Jersey or New York, or be within travel distance to Rutgers University
5. Half of participants will have a best estimate diagnosis of mild to moderate intellectual disability and half will not have intellectual disability. This will be based on participant cognitive assessment and self and/or supporter report of adaptive function during the Baseline visit.

Exclusion Criteria:

1. Are unable to speak and understand English fluently (because the instruments being investigated are currently only validated in English and the focus group and intervention will be delivered in English).
2. Are currently enrolled in another behavioral therapy or psychotherapy targeting depression. Participants will not be excluded if they are currently taking medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change in distress on Patient Health Questionnaire (PHQ-9) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The PHQ-9 is a 9-item self-reported questionnaire of psychological function over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Higher scores equal more distress. The PHQ-9 is administered to those without intellectual disability.
Change in distress on Glasgow Depression Scale (GDS) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The GDS is a 20-item self- and caregiver-reported questionnaire of psychological function over the past week with all items on a "0" (Never/No) to 2 (Always/A lot) scale. Higher scores equal more distress. The GDS is administered to those with intellectual disability.
Change in distress on Anxiety Depression and Mood Scale (ADAMS) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The ADAMS is a 20-item caregiver-reported questionnaire of psychological function over the past week with all items on a "0" (Never/No) to 2 (Always/A lot) scale. Higher scores equal more distress. The ADAMS is administered to those with intellectual disability.
Change on Adult Behavior Checklist (ABCL) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The ABCL is a caregiver-report measure of adaptive functioning and psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true. Higher scores equal more symptoms.
Change on Adult Self Report (ASR) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The ASR is a self-reported measure of adaptive functioning and psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true. Higher scores equal more symptoms.
Change in frequency of activities on Index of Community Involvement (ICI) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The ICI is a 48-item self- and caregiver-reported measure of community involvement over the previous month. All items on the measure ask the frequency of participating in activity from 0 (Never) to 5 (Daily).
Change in frequency of activities on Index of Participation in Domestic Life (IPDL) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The IPDL is an 18-item self- and caregiver-reported measure of participation in domestic activities over the previous month. All items on the measure ask in what manner a participant completed domestic activities from 0 (Did alone without prompting) to 2 (Did not do).
Change in behavioral activation on Behavioral Activation for Depression Scale (BADS) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The BADS is a 25-item self-reported measure of behaviors and thoughts related to depression. All items on the measure ask the participant to rate how much each statement describes them from 0 (not at all) to 6.

SECONDARY OUTCOMES:
Change in adaptive behavior on Vineland Adaptive Behavior Scale, 3rd edition (VABS-3) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The VABS-3 is a 381-item caregiver-reported measure of adaptive behavior. All items in the measure ask the frequency at which the participants performs a behavior, from 0 (never) to 2 (usually).
Change in quality of life on Shalock Quality of Life Questionnaire | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The Shalock Quality of Life Questionnaire is a 40-item self- and caregiver-reported measure of quality of life. Each question prompts the informant to choose one of three options (differing by item) based on which seems most appropriate to them.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa H Bal, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (1):
- Rutgers University - New Brunswick, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No